CLINICAL TRIAL: NCT00645502
Title: A Bioequivalence Study Comparing a Single Oral Intake of a 4mg Orally-disintegrating Tablet With a 4mg Conventional Risperdal Tablet in Patients With Schizophrenia
Brief Title: Bioequivalence Study Comparing 2 Formulations for 4 mg Risperidone Tablet.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR002617
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorders
Keywords: Schizophrenia; Risperidone; Orally-disintegrating tablet; Bioequivalence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The primary objective of this study is to demonstrate the bioequivalence, with respect to risperidone and its active moiety, of a single oral dose of risperidone given as a 4 mg orally-disintegrating tablet and as a 4 mg conventional RISPERDAL tablet. In addition, their tolerability and safety will be documented.

DETAILED DESCRIPTION:
This is a single-center, open, randomized, 2-way crossover bioequivalence study in 40 subjects with schizophrenia or schizoaffective disorder. The study will consist of 2 treatment periods, 5 days per period. The subjects will receive a single 4 mg RISPERDAL conventional tablet in period 1 and a single 4 mg orally-disintegrating tablet in period 2; or the orally disintegrating tablet in period 1 and conventional tablet in period 2. A washout period of at least 10 days between Day 1 of Period 1 and Day 1 of Period 2 will separate the 2 treatments. In both treatment periods plasma concentrations of the drug will be measured. Serial blood collections will be made beginning at 0 hour (immediately before study drug administration) and continuing up to 96 hours after study drug administration in each period. Safety will be evaluated throughout the study using physical examinations, electrocardiogram recordings (ECG), clinical laboratory testing (hematology, serum chemistry, urinalysis), vital signs measurements, pregnancy testing, drug screening, and monitoring of adverse events. The study will be approximately 6 weeks long (including the screening period). Subjects will enter the study facility 3 days before the first administration of study medication on Day 1 of the first period. They will remain at the facility until all study-related procedures are completed on Day 5 of the second study period, a period of approximately 18 days. 4 mg risperidone (either conventional tablet or orally-disintegrating tablet), single dose, oral intake

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of schizophrenia of any subtype
* who have a normal weight as defined by Body Mass Index in range of 18.0 to 35.0, extremes included
* For whom an Informed consent form signed by the patient or legally acceptable representative is available and who are healthy on the basis of a pre-trial physical examination, medical history, electrocardiogram (ECG), and the results of blood biochemistry and hematology tests and a urinalysis carried out less than 3 weeks before the first dose of study medication is taken

Exclusion Criteria:

* Patients with a mental disorders other than schizophrenia or schizoaffective disorder, according to the DSM-IV
* Patients who received oral risperidone or paliperidone within 14 days of first drug administration, Risperdal Consta within 100 days of first drug administration or paliperidone palmitate within 10 months of first drug administration
* Patients who used medication known to be an hepatic enzyme inducer or inhibitor less than 2 weeks prior to first drug administration
* Patients with history of allergic reaction to risperidone or its excipients
* Patients with diagnosis of alcohol or substance abuse
* Patients with history of clinically relevant cardiac arrhythmia's, bronchospastic or cardiovascular disease, diabetes mellitus, thyrotoxicosis, parkinsonism, or drug allergy
* Female patients who are pregnant or are breastfeeding or are of childbearing potential without adequate contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-06; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
PK parameters (Cmax and AUC) for active moiety, 9-OH-risperidone and risperidone

SECONDARY OUTCOMES:
Safety assessments including adverse events, physical examination, vital signs, ECGs and labs

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.